CLINICAL TRIAL: NCT05793177
Title: Monitoring Sedentary Behavior and Light Physical Activity in Patients With Stroke
Acronym: MONSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Sjørslev Bodilsen, Ph.d. student, MSPT, PT, Zealand University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MONSS
Record Dates: First submitted 2023-03-23; First posted 2023-03-31 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Acute; Behavior; Physical Inactivity; Sedentary Behavior
MeSH Terms: conditions — Stroke; Behavior; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Everyday Life is Rehabilitation
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Everyday Life is Rehabilitation — Behavior change intervention focuses on implementing more movement into everyday life using action planning, goal setting, and fatigue management.
  Arms: Intervention

SUMMARY:
This randomized control trial (RCT) aims to test the effect of a 12 weeks tailored behavioral intervention on stroke survivors living in the community and compare the results to a control group of stroke survivors participating in standard care. The intervention's purpose is to lower the time spend with sedentary behavior and raise the level of physical activity in stroke survivors throughout their everyday life. The intervention contains two motivational interviews with a focus on goal setting, action planning, motivation, fatigue management, and general information on life after stroke. The primary outcome for behavior change is objectively measured physical activity using an activity tracker (ActivPal4 Micro) and secondary glycohemoglobin and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Verified ischemic stroke or intracerebral hemorrhage
* Modified rankin score (mRS) 1-3 at discharge
* Discharged with at rehabilitation plan within 1-14 hospitalization days
* Able to ambulate independently
* Speak and understand Danish

Exclusion Criteria:

* Aphasia
* Unable to give informed consent
* Unable to ambulate independently
* Mental illness
* Other co-morbidity like terminal cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sedentary time | 12 weeks follow-up
  Time participants spend with sedentary behavior compared between the intervention and control group

SECONDARY OUTCOMES:
Physical activity scale (PAS2) | Baseline,12 and 26 weeks follow-up
  Subjective physical activity
The Stroke Specific Quality of Life Scale (SS-QOL) | Baseline,12 and 26 weeks follow-up
  Quality of life
The General Self-efficacy Scale (GSES) | Baseline,12 and 26 weeks follow-up
  self-efficacy
The Multi-dimensional Fatigue Inventory (MFI-20) questionnaire | Baseline,12 and 26 weeks follow-up
  Fatigue
Patient health questionnaire (PHQ-9) | Baseline,12 and 26 weeks follow-up
  Depression symptoms
The Fugl Meyer Assessment (FMA) | Baseline,12 and 26 weeks follow-up
  The function of upper and lower extremity
Timed Up & Go (TUG) test | Baseline,12 and 26 weeks follow-up
  Mobility
Montreal Cognitive Assessment (MoCA) | Baseline
  cognitive assessment
Glycated hemoglobin (HbA1c) | Baseline,6,12 and 26 weeks follow-up
  Glycated hemoglobin (HbA1c)

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University hospital, Roskilde, Denmark

REFERENCES:
- [Background] Bodilsen SS, Aadahl M, Wienecke T, Thomsen TH. Development of a tailored intervention targeting sedentary behavior and physical activity in people with stroke and diabetes: A qualitative study using a co-creation framework. Front Rehabil Sci. 2023 Feb 13;4:1114537. doi: 10.3389/fresc.2023.1114537. eCollection 2023. PMID 36860816